CLINICAL TRIAL: NCT04927338
Title: Phase II, Placebo-controlled Study of BacoMind® Bacopa Monnieri Standardized Extract in Gulf War Illness
Brief Title: Study of Bacopa in Gulf War Illness Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: RTI International (Other); Boston University (Other)
Responsible Party: Principal Investigator, Amanpreet Cheema, Assistant Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWICTIC-Bacopa; W81XWH1820062 (Other Grant/Funding Number: US DoD USAMRAA)
Record Dates: First submitted 2021-06-07; First posted 2021-06-16 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Gulf War Illness
Keywords: Veterans; Gulf War Illness; Nutraceutical

STUDY DESIGN:
Intervention Model Description: This is a double-blinded, two-arm, placebo-controlled, randomized phase II study in 170 participants born between 1946 and 1978 who are Gulf War Veterans and meet the modified Kansas and Centers for Disease Control and Prevention (CDC) case definition for Gulf War Illness.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care providers, investigators, study coordinators, and laboratory technicians will be masked to the participants' treatment group status. Placebo capsules will be identical in size, color, and shape to that of the Bacopa capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BacoMind® 300mg/day (Experimental): Participants randomized to the experimental arm will receive 12 weeks of 300 mg/day BacoMind® Bacopa monnieri standardized extract.
  Interventions: Dietary Supplement: BacoMind® (Bacopa monnieri standardized extract)
- Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive 12 weeks of daily placebo identical to the experimental treatment in size, color, and shape.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: BacoMind® (Bacopa monnieri standardized extract) — BacoMind® (Bacopa monnieri standardized extract) 300 mg daily capsule.
  Other Names: Bacopa; Bacopa monnieri
  Arms: BacoMind® 300mg/day
Drug: Placebo — Daily placebo capsule identical in size, color, and shape to that of the Bacopa capsules.
  Arms: Placebo

SUMMARY:
Gulf War Illness is a condition that affects multiple major organ systems, resulting in a diverse array of symptoms that include debilitating fatigue, memory and cognition difficulties, headaches, sleep disturbances, gastrointestinal problems, skin rashes, and musculoskeletal/joint pain. This phase II, double masked, randomized, placebo-controlled, two-arm study will evaluate cognitive function as evidence of efficacy of the nutraceutical intervention, Bacopa, on central nervous system symptom management of Gulf War Illness, along with assessments of safety of the intervention.

DETAILED DESCRIPTION:
This is a study in Gulf War Veterans born between 1946 and 1978 who meet the modified Kansas and Centers for Disease Control and Prevention (CDC) case definitions for Gulf War Illness. This phase II, double-masked, randomized, placebo-controlled, two-arm study will focus on assessing cognitive function as evidence of efficacy of the nutraceutical intervention, Bacopa, on central nervous system symptom management of Gulf War Illness. 170 participants will be randomized 1:1 to receive either 12 weeks of the intervention (Bacopa) or placebo. Participants will be evaluated "remotely" via online assessment tools and telephone interviews, allowing participation from a nationwide catchment area. Primary assessment via the California Verbal Learning Test, Second Edition (CVLT-II) will occur at baseline and 12 weeks, along with laboratory assessments for all participants at baseline, and a self-selected subgroup at 12 weeks. Randomization to the intervention or placebo arms will be stratified by membership in the 12-week follow-up laboratory subgroup and sex. Laboratory draws will be performed at the participant's local clinical laboratory and will allow for measurements of putative biomarkers of neuron health and structural integrity along with biomarkers of inflammation and immune signaling. Monitoring phone calls will be made to the participant biweekly to assess safety. Participants will also undergo subjective assessments of physical health, vitality, sleep, pain, and symptom severity at baseline, 6, 12, and 16 weeks. Thus, participants will be observed through the treatment period (12 weeks) and for 4 weeks after completion to assess immediate effects and durability of the response.

ELIGIBILITY:
Inclusion Criteria:

1. Born in years 1942 to1978
2. Served in the Gulf War theater for any period between August 1990 and July 1991
3. Meets modified Kansas case definition criteria and CDC case definition for Gulf War Illness (GWI). The modified Kansas definition, which includes the CDC criteria includes:

   1. Allowance for normal illnesses of aging, such as hypertension and diabetes if the conditions are treated and are in demonstrable stable and normal ranges at the time of screening and assessment.
   2. Allowance of stable comorbid conditions such as post-traumatic stress disorder (PTSD), major depressive disorder (MDD), and traumatic brain injury (TBI) that have not required hospitalization in the 5 years prior to recruitment. Severe TBI is excluded.
4. Able to consent to the study
5. Participants of childbearing potential must practice effective contraception during the study so that, in the opinion of the Investigator, they will be compliant with birth control measures during the study.
6. Agrees to participate in follow-up visits.

Exclusion Criteria:

1. They are scheduled for a surgery during the period of study participation, had minor surgery within 3 months prior to screening, or had major surgery within 6 months prior to screening,
2. Self-report of current untreated major depression with psychotic or melancholic features (as determined by self-report), schizophrenia, bipolar disorder, delusional disorders, dementias of any type, or substance abuse during the last two years (excluding cannabis products),
3. Any serious allergic disease (self-report), possibly resulting in anaphylaxis, such as food/drug allergies, including allergic asthma, or allergy to any ingredient of the active product or placebo, including allergies to FD&C Yellow No. 5 (tartrazine),
4. Renal disease (self-report; laboratory results: renal insufficiency with serum creatinine > 2.0 mg/dL or eGFR < 44; or currently on renal dialysis),
5. Hepatic insufficiency (bilirubin >2.5mg/dL or transaminases >3x the upper limit of normal (ULN)). Participants with Gilberts syndrome are eligible for the study if other liver function tests are normal, regardless of bilirubin level,
6. Pregnancy (premenopausal female participants),
7. Current heavy alcohol or tobacco use (self-report). Heavy use is defined as alcohol consumption not to exceed approximately 15 drinks per week (with a drink defined as 12 oz beer, 5 oz wine, or 1.5 oz distilled spirits) and tobacco use not to exceed 20 cigarettes (or equivalent) per day.
8. Current exclusionary diagnosis that could reasonably explain the symptoms of their fatiguing illness and their severity, using the exclusion criteria best described in the Ambiguities in case definition paper for Chronic Fatigue Syndrome (CFS), as described in detail in Reeves et al., 2003, which clarifies exclusionary conditions. Specifically, the exclusionary diagnoses that are not otherwise listed above comprise:

   * organ failure (e.g., emphysema, cirrhosis, cardiac failure, chronic renal failure)
   * chronic infections (e.g., AIDS, hepatitis B or C) or inflammatory bowel disease (IBD) (via self report)
   * major neurologic diseases that could cause fatigue or neurologic deficits such as (e.g., epilepsy, stroke, brain tumor, multiple sclerosis, Parkinson's Disease, Alzheimer's disease) or history of CNS demyelinating disease (e.g., multiple sclerosis, neuromyelitis optica spectrum disorder) (Self report),
   * cancer or cancer treatment (e.g., chemotherapy, radiation of brain), or current use of biologic modifiers that could affect immune function (e.g., Etanercept, Rituximab) (self-report)
   * untreated primary sleep disorders (e.g., sleep apnea, narcolepsy)
   * uncontrolled diabetes (HgbA1c > 7)
9. Temporary conditions discovered at screening for which participants may be rescreened 6 weeks after resolution of condition.

   * Temporary effects of medications
   * Temporary sleep deprivation
   * Untreated hypothyroidism/hyperthyroidism, hypothyroidism/hyperthyroidism that has been inadequately controlled during the last 3 months, or free T4 level not within normal limit
   * Active infection
10. Participating in another interventional clinical trial of an investigational therapy (including social-behavioral therapy) within 6 weeks prior to consent to participate in this study, or planning to participate in another interventional clinical trial of an investigational therapy during this study,
11. Use of Bacopa within 6 weeks prior to the enrollment in this study,
12. Diagnosed bleeding disorder or current use of anticoagulants and/or antiplatelets, except for low dose nonsteroidal anti-inflammatories (NSAIDS).

Ages: 46 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
California Verbal Learning Test (CVLT-II) Assessment | 12 weeks
  Change in mean CVLT-II long delay free recall from baseline to 12 weeks. Higher CVLT-II scores are considered clinically better, and the raw CVLT-II scores will be used in analyses and reporting.

SECONDARY OUTCOMES:
Blood Biomarker Concentrations | 12 weeks
  Putative biomarkers 18-plex cytokines, glutamate, brain-derived neurotrophic factor (BDNF), and neurofilament light chain (NfL) will be measured from blood drawn at baseline from all participants and then at 12 weeks from a subgroup of participants. Differences in the mean concentrations of each of the biomarkers will be assessed at the end of the intervention period in the 12 week blood draw subgroup.
Veterans RAND 36 Item Health Survey (VR-36©) | 12 weeks
  Change in mean VR-36 physical component score from baseline to 12 weeks. Normed values of the VR-36 physical component score (PCS) will be used based on US population estimates. The minimum score is 0 and the maximum score is 100. A higher score indicates better health outcomes.
Veterans RAND 36 Item Health Survey (VR-36©) | 16 weeks
  Change in mean VR-36 physical component score (PCS) from 12 weeks to 16 weeks. Normed values of the VR-36 PCS will be used based on US population estimates. The minimum score is 0 and the maximum score is 100. A higher score indicates better health outcomes.
Review of Treatment Related Adverse Events | 16 weeks
  Number of participants with treatment-related adverse events as assessed by frequency of safety events during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Amanpreet Cheema, PhD, Principal Investigator — Nova Southeastern Univeristy
Locations (1):
- Nova Southeastern University, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The plan is to release primary results from the study to ClinicalTrials.gov. Data are the property of Nova Southeastern University, but data and publication thereof will not be unduly withheld. Those interested in Bacopa data should reach out to Amanpreet Cheema (PI) for more information.